CLINICAL TRIAL: NCT05288530
Title: Satisfaction, Pain and Function Outcomes of Breast Reduction Patients: A Retrospective Chart Review and Patient Follow up
Brief Title: Satisfaction, Pain and Function Outcomes of Breast Reduction Patients
Status: Completed | Type: Observational
Sponsor: Claytor Noone Plastic Surgery (Other)
Responsible Party: Sponsor
Other Study IDs: R17-3683B
Record Dates: First submitted 2021-08-02; First posted 2022-03-21 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Macromastia; Hypertrophy Breast
MeSH Terms: conditions — Gigantomastia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To explore the indications and benefits of breast reduction. The investigators suspect all of the patients in this population suffer from neck/back pain and limitations in function. The investigators also want to review the patients in this group to determine if the amount of breast tissue removed or previous breast size affects outcomes for these patients. Patients will then be contacted for outcome data and satisfaction information. Ultimately, this information may lead to improvements in management and education of patients with macromastia.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Ages 21-71 years-old
* Hypertropy of the breast
* Macromastia
* post-surgical intervention for macromastia or hypertrophy of the breast

Exclusion Criteria:

* Males
* BMI>40
* Hypertrophy of the breast but without surgical intervention
* Macromastia but without surgical intervention

Ages: 21 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients between the age of 21-70 diagnosed with hypertrophy of the breast or macromastia with surgical intervention
Study Population: Females age 21-70 with a diagnosis of hypertrophy of the breast who underwent surgical intervention
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
DASH questionnaire | 6 months
  Disabilities of the arm shoulder and hand, pain and function indicators
Breast Q questionnaire | 6 months
  quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Brannon Claytor, Principal Investigator — Claytor Noone Plastic Surgery